CLINICAL TRIAL: NCT06898918
Title: Association Between Maternal Control of the Child's Feeding, Child's Eating Behavior and Early Childhood Caries in Preschoolers: A Cross-Sectional Study
Brief Title: Maternal Control of the Child's Feeding, Child's Eating Behavior and Early Childhood Caries in Preschoolers
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ayman Amin Sharaf, Assistant lecturer of dental public health, Ain Shams University
Other Study IDs: 1315
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries in Children; Diet Habit; Dietary Exposure; Eating Behavior; Parent-Child Relations; Body Weight
MeSH Terms: conditions — Feeding Behavior; Body Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dental caries in children is considered one of the most prevalent oral diseases of this age group, leading to significant manifestations presenting as pain, interference with feeding, higher risk of developing dental caries in both, primary and permanent dentition. Dietary practices, along with the presence of bacteria in the oral cavity have been shown to be inextricably linked to the presence of dental caries. The latest evidence has demonstrated that certain types of eating behavioral traits in children could influence the development of dental caries.

DETAILED DESCRIPTION:
Dental caries in children is considered one of the most prevalent oral diseases of this age group, leading to significant manifestations presenting as pain, interference with feeding, higher risk of developing dental caries in both, primary and permanent dentition, as well as worse repercussions on the permanent successors. According to the World Health Organization (WHO) global oral health status report of 2022, 514 million children -worldwide- have been affected by dental caries in their primary teeth. The American Academy of Pediatric Dentistry (AAPD) refers to this type of dental caries in primary teeth as "early childhood caries" and defines it as the existence of one or more decayed, missed, or filled tooth surface due to dental caries in children less than six years of age.

It has been studied in depth that dental caries is a multi-factorial disease of a complex nature with behavioral, as well as social factors playing a vital role in its etiology. Dietary practices, along with the presence of bacteria in the oral cavity have been shown to be inextricably linked to the presence of dental caries. The latest evidence has demonstrated that certain types of eating behavioral traits in children could, in a way, influence the development of dental caries.

Moreover, family structure could be an additional, recently confirmed factor to contemplate in regards to the etiology of dental caries. For example, it has been shown that parents, as the primary caregiver of the child, could influence the eating habits of their preschool children. This could occur through parents choosing the food they consider "appropriate" for their child, modelling, creating specific patterns of feeding for the child and adopting particular food practices to reinforce eating behaviors in their children.

Several questionnaires that assess the child's eating behavioral traits as well as parental control of the child's feeding have been found in the literature, among which, the most frequently used are the "Children's Eating Behavior Questionnaire (CEBQ)" and the "Child Feeding Questionnaire (CFQ)". Both questionnaires have been shown to have good psychometric properties and both have been validated and translated to Arabic language in recent studies.

Research suggests that evidence on the relationship between children's eating behavior and dental caries is scanty. Additionally, the association between parental control in child feeding and dental caries has been investigated in a limited number of studies. To our knowledge, to date, this type of research has not been previously conducted in Egypt. On that account, this study has been developed with the aim of investigating the relationship between parental control in child feeding, child's eating behavior and dental caries in a number of Egyptian preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian mothers and preschool children pairs aging from 3-5 years old, and currently residing in Egypt.
* Mothers who live with the child in the same household

Exclusion Criteria:

* Participants who refuse to consent to participate in the study.
* Mothers with any medical health condition (physical or mental) that interferes with responding to the questionnaires.
* Children with special health care needs (mental or physical).
* Medically compromised children (Diabetic, renal problems, liver problems, respiratory problems…etc.) as their condition or the medications they consume might interfere with their oral health status.
* Children whose siblings have previously participated in the study.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother-child pairs attending the Faculty of Dentistry, Ain Shams University will be recruited and enrolled in the current study
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Early childhood caries | January 2025 - June 2026
  Early childhood caries will be assessed using decayed, missing, and filled tooth index (dmft)

SECONDARY OUTCOMES:
Oral hygiene condition (oral debris) | January 2025 - March 2027
  The Debris Index-Simplified (DI-S), a component of the Oral Hygiene Index-Simplified (OHI-S) by Silness and Loe will be used to evaluate the oral hygiene of children.
  - Six index teeth will be assessed to obtain a final score: The labial/buccal surface of the primary maxillary right central incisor, primary mandibular left central incisor, primary maxillary right second molar, and primary maxillary left second molar. Whereas the lingual surface of the primary mandibular left and right second molar will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Badran, PhD, Study Director — Ain Shams University; Nagwa Khattab, PhD, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonotto DV, Montes GR, Ferreira FM, Assuncao LRDS, Fraiz FC. Association of parental attitudes at mealtime and snack limits with the prevalence of untreated dental caries among preschool children. Appetite. 2017 Jan 1;108:450-455. doi: 10.1016/j.appet.2016.11.007. Epub 2016 Nov 3. PMID 27818303
- [Background] Mosli RH. Validation of the Child Feeding Questionnaire among Saudi pre-schoolers in Jeddah city. Public Health Nutr. 2020 Mar;23(4):599-608. doi: 10.1017/S1368980019002581. Epub 2019 Sep 13. PMID 31516100
- [Background] Shqair AQ, Dos Santos Motta JV, da Silva RA, do Amaral PL, Goettems ML. Children's eating behaviour traits and dental caries. J Public Health Dent. 2022 Mar;82(2):186-193. doi: 10.1111/jphd.12449. Epub 2021 Mar 15. PMID 33719035
- [Background] Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. Appetite. 2001 Jun;36(3):201-10. doi: 10.1006/appe.2001.0398. PMID 11358344
- [Background] Al-Hamad AH, Al-Naseeb AM, Al-Assaf MS, Al-Obaid SA, Al-Abdulkarim BS, Olszewski PK. Preliminary Exploration of Obesity-Related Eating Behaviour Patterns in a Sample of Saudi Preschoolers Aged 2-6 Years through the Children's Eating Behaviour Questionnaire. Nutrients. 2021 Nov 20;13(11):4156. doi: 10.3390/nu13114156. PMID 34836411